CLINICAL TRIAL: NCT00006120
Title: Phase II Randomized Study of Two Different Schedules of Docetaxel or Paclitaxel for Metastatic Breast Cancer
Brief Title: Docetaxel or Paclitaxel in Treating Women With Unresectable Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068134; FRE-GERCOR-TAXMAX-SOO-1; EU-20029
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2006-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Paclitaxel

INTERVENTIONS:
Drug: docetaxel
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to compare the effectiveness of two different regimens of docetaxel or paclitaxel in treating women who have unresectable locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rate, progression free survival, and overall survival in women with unresectable locally advanced or metastatic breast cancer treated with two different schedules of docetaxel or paclitaxel.
* Compare the toxicities and pharmacoeconomics of these four regimens in these patients.
* Compare the quality of life of patients treated with these four regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center, age, ECOG performance status, hormone receptor status (positive vs negative), metastasis to liver (yes vs no), and presence of disease progression following anthracyclines (yes vs no).

Patients are randomized to one of four treatment arms.

* Arm I: Patients receive docetaxel IV over 1 hour on day 1.
* Arm II: Patients receive paclitaxel IV over 3 hours on day 1.
* Arm III: Patients receive docetaxel IV over 1 hour on days 1, 8, 15, 22, 29, and 36.
* Arm IV: Patients receive paclitaxel IV over 1 hour on days 1, 8, 15, 22, 29, and 36.

Courses repeat every 3 weeks (arms I and II) or every 8 weeks (arms III and IV) in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed prior to treatment and then every 8 weeks.

PROJECTED ACCRUAL: A total of 165 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven unresectable locally advanced or metastatic breast cancer

  * Refractory or relapsed disease after neoadjuvant or adjuvant anthracyclines
* At least one bidimensionally measurable lesion
* No brain metastasis
* No bone metastases, lymphangitis carcinomatous, ascites, or pleural effusion as sole site of metastatic disease
* Hormone receptor status:

  * Known hormone receptor status

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* AST and ALT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* Bilirubin normal

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled angina or arrhythmia
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart disease

Other:

* No sensitive neuropathy worse than grade 2
* No other significant, uncontrolled medical or psychiatric condition
* No serious active infection
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other prior malignancy except treated nonmelanomatous skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior specific antitumoral immunotherapy

Chemotherapy:

* See Disease Characteristics
* No prior taxanes
* At least 4 weeks since other prior specific antitumoral chemotherapy

Endocrine therapy:

* At least 4 weeks since prior specific antitumoral hormonal therapy

Radiotherapy:

* At least 4 weeks since prior specific antitumoral radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent experimental medication

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gligorov, MD, Study Chair — Hopital Tenon
Locations (35):
- France (34):
  - Centre Hospitalier d'Antibes, Antibes
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Institut Sainte Catherine, Avignon
  - Clinique Floreal, Bagnolet
  - Centre D'Oncologie Du Pays-Basque, Bayonne
  - C.H.G. Beauvais, Beauvais
  - Hopital Fontenoy, Chartres
  - Centre Jean Perrin, Clermont-Ferrand
  - Hopital Louis Mourier, Colombes
  - Centre Hospitalier Laennec, Creil
  - Hopital Intercommunal De Creteil, Créteil
  - Hopital Drevon, Dijon
  - Polyclinique Jeanne d'Arc - service de Radiotherapie Oncologie, Gien
  - Centre Jean Bernard, Le Mans
  - Hopital Desgenettes - Service de Medecine Interne, Lyon
  - Centre de Radiotherapie et Oncologie Saint-Faron, Mareuil-lès-Meaux
  - Hopital Saint Joseph, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - CH Meulan, Meulan-en-Yvelines
  - Intercommunal Hospital, Montfermeil
  - Centre Hospitalier de Mulhouse, Mulhouse
  - Clinique Hartmann, Neuilly-sur-Seine
  - American Hospital of Paris, Neuilly-sur-Seine
  - Clinique Geoffroy St. Hillaire, Paris
  - Hotel Dieu de Paris, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Clinique Ste - Marie, Pontoise
  - Polyclinique De Courlancy, Reims
  - Centre du Rouget, Sarcelles
  - C.H. Senlis, Senlis
  - Clinique de l'Orangerie, Strasbourg
  - Clinique Pasteur, Toulouse
  - Clinique Fleming, Tours
- Hopital de la Ville D'Esch-sur-Alzette, Esch-sur-Alzette, Luxembourg